CLINICAL TRIAL: NCT06364098
Title: Comparative Study Between the Roles of Intrauterine Misoprostol Versus the Sublingual Route for Prevention of Postpartum Blood Loss in Elective Cesarean Sections: A Randomized Controlled Trial
Brief Title: Comparative Study Between the Roles of Intrauterine Misoprostol Versus the Sublingual Route for Prevention of Postpartum Blood Loss in Elective Cesarean Sections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adel Atef, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: prevention of PPH
Record Dates: First submitted 2024-03-24; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intrauterine misoprostol group (Group A) (Experimental): 96 women receiving 400 mcg intrauterine misoprostol + IV oxytocin.
  Interventions: Drug: Misoprostol
- sublingual misoprostol group (Group B) (Active Comparator): : 96 women receiving 400 mcg sublingual misoprostol + IV oxytocin.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400 microgram of misoprostol given either sublingually or intrauterine during CS after placental removal together with IV oxytocin infusion

SUMMARY:
Study design:

A prospective randomized control trial was carried out at labor and delivery unit at Kasr Al Aini Hospital, Cairo University.

Population of study:

192 pregnant women at the age range from 20 to 35 years, with BMI < 30kg/m2 presenting with a full-term singleton healthy living fetus (gestational age >39 weeks confirmed by the first day of the last menstrual period or first-trimester ultrasound scan) and candidate for elective cesarean delivery (Previous one or two cesarean section) were included in our study. Patients with uterine over distension as due to multiple pregnancies or polyhydramnios, multipara (parity ≥3), women with uterine fibroids, antepartum hemorrhage presentation such as placenta previa, placental abruption or vasa previa, moderate to severe anemia with hemoglobin level <9mg/dl, patient on anticoagulant during pregnancy or having coagulopathy or thrombocytopenia or blood dyscrasias, hypertension, cardiovascular, DM, hepatic, or renal disorders and women with any contraindication for the use of misoprostol or oxytocin as allergy to prostaglandin and concomitant drugs that have drug interaction with prostaglandins as topical dinoprostone, antacids containing magnesium were excluded from our study.

DETAILED DESCRIPTION:
After receiving the research approval of the Scientific and Ethical Committee of the Obstetrics and Gynecology department, Cairo University, the study purpose was clarified simply and in a lay Arabic speech to all women before registering in the study, and the enrolled women signed informed consent form. Pregnant women who met all the inclusion criteria were evaluated for enrollment. Prior to the study, randomization schedules created by computer program were designed and settled in serially numbered secured opaque envelopes. Simple randomization was applied at one to one ratio within both groups. The recruited women - after giving consent for participation- opened the sealed randomization envelopes for revealing the allocation.

All participants were subjected to Comprehensive history taking including obstetric, medical, and surgical history.

General examination excluding the presence of any abnormalities. Systematic obstetrical examinations. A transabdominal ultrasound to confirm the diagnosis and evaluation of fetal condition.

A blood sample collected for complete blood counting, coagulation studies, liver and kidney function tests.

All women were subjected to elective lower segment cesarean section by the same team under spinal anesthesia and antibiotic prophylaxis according hospital protocol.

Women were divided into two equal groups:

Group A: 96 women receiving 400 mcg intrauterine misoprostol + IV oxytocin. Group B: 96 women receiving 400 mcg sublingual misoprostol + IV oxytocin. Both groups were subjected to the same preparation. All cesarean deliveries were performed by a senior obstetrics and gynecology resident and the elective sections were performed at 39th weeks gestation adopting the following operative steps: transverse skin incision (Pfannenstiel), smiley incision at the lower uterine segment, immediate clamping of the cord within 30 seconds, placental extraction after its spontaneous separation, two layers closure of the uterine incision, and abdominal closure anatomically in layers. All surgical steps were done with adequate hemostasis. Furthermore, the investigators excluded sections exceeding 90 minutes from skin incision to skin closure.

After fetal head extraction, participants in both groups were given 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) as intravenous bolus and continued on infusion of 10 IU oxytocin in 500 mL of Ringer lactate at a rate of 125 mL/hour.

* For all women in group A: the surgeon placed two intrauterine misoprostol tablets (Misotac® 200microgram, Sigma Ph., Egypt) at the fundus after placental delivery and swabbing the cavity followed by suturing the first layer of the uterus, while women in group B were given two sublingual misoprostol tablets (Misotac® 200 microgram, Sigma Ph., Egypt) after placental delivery.
* The amount of blood loss was determined through the standardized visual estimation method and rectified by measuring the amount of intraoperative blood loss and 6 hours after surgery. The estimated total blood loss during cesarean section was measured after adding the volume of blood in the suction bottle to the soaked surgical towels (weighting method) then added to the amount of blood lost after section calculated by using blood collection drape. Moreover, hemoglobin (HB) level and hematocrit value were repeated 24 hours postpartum. The patient vitals were observed and recorded intraoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-35 years.
2. BMI < 30kg/m2.
3. Singleton pregnancy.
4. Full term pregnancies (recruiting from 37 weeks of gestation).
5. Elective cesarean section (previous one or two cesarean section).

Exclusion Criteria:

1. Active labour before 39 weeks.
2. Uterine over distension as due to multiple pregnancies or polyhydramnios.
3. Multipara [parity ≥3].
4. Pregnancy with obstetric haemorrhage such as placenta Previa, placental abruption or vasa Previa.
5. Moderate to severe anemia with HB <9mg/dL.
6. Pregnancy with coagulopathy, thrombocytopenia or blood dyscrasias.
7. Women with uterine fibroids.
8. Medically complicated pregnancy (pregnancy induced hypertension, cardiovascular, DM, hepatic, or renal disorders).
9. Women with any contraindication for the use of misoprostol or oxytocin as a history of prostaglandin allergy and current medication which could cause severe drug interaction to prostaglandins such as topical dinoprostone, magnesium-containing antacids or quinapril.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The amount of blood loss | 6 hours
  determined through the standardized visual estimation method and rectified by measuring the amount of intraoperative blood loss and 6 hours after surgery

SECONDARY OUTCOMES:
Changes in hematocrit values in both groups after delivery | 24 hours
  Hematocrit values measured before section and 24 hours after section
Changes in Hemoglobin level measured by gm/dl in both groups after delivery | 24 hours
  Hemoglobin level in gm/dl measured before section and 24 hours after section

OTHER OUTCOMES:
Incidence of side effects of study medications | 24 hours
  shivering, pyrexia >38°C, headache, nausea, vomiting with or without the need for anti-emetic drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Kasr Alainy, Cairo, Al Manyal, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gallos I, Williams H, Price M, Pickering K, Merriel A, Tobias A, Lissauer D, Gee H, Tuncalp O, Gyte G, Moorthy V, Roberts T, Deeks J, Hofmeyr J, Gulmezoglu M, Coomarasamy A. Uterotonic drugs to prevent postpartum haemorrhage: a network meta-analysis. Health Technol Assess. 2019 Feb;23(9):1-356. doi: 10.3310/hta23090. PMID 30821683
- [Background] Gallos ID, Williams HM, Price MJ, Merriel A, Gee H, Lissauer D, Moorthy V, Tobias A, Deeks JJ, Widmer M, Tuncalp O, Gulmezoglu AM, Hofmeyr GJ, Coomarasamy A. Uterotonic agents for preventing postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2018 Apr 25;4(4):CD011689. doi: 10.1002/14651858.CD011689.pub2. PMID 29693726
- [Background] Escobar MF, Nassar AH, Theron G, Barnea ER, Nicholson W, Ramasauskaite D, Lloyd I, Chandraharan E, Miller S, Burke T, Ossanan G, Andres Carvajal J, Ramos I, Hincapie MA, Loaiza S, Nasner D; FIGO Safe Motherhood and Newborn Health Committee. FIGO recommendations on the management of postpartum hemorrhage 2022. Int J Gynaecol Obstet. 2022 Mar;157 Suppl 1(Suppl 1):3-50. doi: 10.1002/ijgo.14116. No abstract available. PMID 35297039
- [Background] Awoleke JO, Adeyanju BT, Adeniyi A, Aduloju OP, Olofinbiyi BA. Randomised Controlled Trial of Sublingual and Rectal Misoprostol in the Prevention of Primary Postpartum Haemorrhage in a Resource-Limited Community. J Obstet Gynaecol India. 2020 Dec;70(6):462-470. doi: 10.1007/s13224-020-01338-0. Epub 2020 Jun 29. PMID 33417650
- [Background] Bagheri FZ, Azadehrah M, Shabankhani B, Nasiri Formi E, Akbari H. Rectal vs. sublingual misoprostol in cesarean section: Three-arm, randomized clinical trial. Caspian J Intern Med. 2022 Winter;13(1):84-89. doi: 10.22088/cjim.13.1.84. PMID 35178212
- [Derived] Atef A, Shehata HSEAM, Bassiouny YA, Al-Inany HG. Comparative study between the roles of intrauterine misoprostol versus the sublingual route for prevention of postpartum blood loss in elective cesarean sections: a randomized controlled trial. BMC Pregnancy Childbirth. 2024 Oct 29;24(1):710. doi: 10.1186/s12884-024-06889-y. PMID 39472831